CLINICAL TRIAL: NCT07405099
Title: The Analysis of End-stage Renal Disease for Outcomes in Pancreatic Surgery
Brief Title: Operative Risk After Pancreatic Surgery in Patients With End Stage Renal Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Clinical Professor, National Taiwan University Hospital
Other Study IDs: 202107127RINB
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Neoplasms
Keywords: pancreatic surgery; end-stage renal disease; renal placement therapy
MeSH Terms: conditions — Pancreatic Neoplasms; Kidney Failure, Chronic | interventions — Pancreatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pancreatectomy — Any operation demanding pancreatic parenchyma transaction

SUMMARY:
End-stage renal disease (ESRD) patients often present risk factors for many surgical complications. The severity of renal failure and whether the patient is receiving renal replacement therapy are also related to the difficulty of pancreatic and other major surgeries, causing many ESRD patients to hesitate when choosing surgery. Therefore, this project aims to retrospectively collect basic data, preoperative and postoperative blood tests (blood cell counts, biochemistry, tumor markers, glucose-related, lipid-related), and preoperative and postoperative imaging examinations (CT, MRI, Ultrasound, PET scan, Endoscopy, etc.) of ESRD patients who underwent pancreatic surgery at our hospital. We aim to compare whether surgical methods, severity of renal failure, use of renal replacement therapy, and lesion margin clearance rates affect the occurrence of surgical complications, length of hospital stay, length of ICU stay, re-operation rates or severe complications, medical costs, and related quality of life. This analysis is intended to understand and analyze the surgical prognosis, care priorities, common complications, and the management and outcomes of our team for ESRD patients undergoing pancreatic surgery, with the expectation of providing more diverse and specific treatment recommendations for these patients in the future.

DETAILED DESCRIPTION:
Background End-stage renal disease patients often present risk factors for many surgical complications. However, the severity of renal failure and whether the patient is receiving renal replacement therapy are also related to the difficulty of pancreatic and other major surgeries, causing many end-stage renal disease patients to hesitate when choosing surgery options.

IV. Objectives To compare whether surgical methods, severity of renal failure, use of renal replacement therapy, and lesion margin clearance rates affect the patient's occurrence of surgical complications, length of hospital stay, length of ICU stay, re-operation or severe complications, medical costs, and related quality of life.

V. Methodology and Procedures Data Collection The Principal Investigator and Co-Investigator will retrospectively review medical records to collect basic data of patients with end-stage renal disease who underwent pancreatic surgery at this hospital. This includes preoperative and postoperative blood tests (blood counts, biochemistry, tumor markers, glucose-related, lipid-related) and imaging examinations (CT, MRI, Ultrasound, PET scan, Endoscopy, etc.). This data will be used to compare the impact of surgical methods, renal failure severity, renal replacement therapy status, and margin clearance on surgical complications, hospital stay, ICU stay, re-operations, severe complications, medical costs, and quality of life. The goal is to analyze the prognosis, care priorities, and management outcomes for ESRD patients undergoing pancreatic surgery.

From the hospital portal system, approximately 500 medical records of patients with pancreatic diseases who underwent pancreatic surgery or invasive treatment performed by the Principal Investigator and Co-Investigator between January 2005 and July 2021 will be collected. This observational study will collect routine imaging and laboratory tests performed at the hospital to analyze treatment indications, surgical indicators, and prognosis.

Inclusion Criteria:

1. Males or females aged 20 years or older.
2. Patients scheduled to undergo pancreatic surgery.

Exclusion Criteria:

1. Patients under 20 years of age at this hospital.
2. Presence of other active malignancies prior to diagnosis.
3. Minors, pregnant women, breastfeeding women, and patients with psychiatric disorders.

Treatment Flow For patients after pancreatic surgery, daily records will be kept regarding vital signs, drainage volume, intake/output balance, dietary intake and emptying, occurrence/management/severity of complications, length of hospital stay, length of ICU stay, re-operations or severe complications, medical costs, related quality of life, and nutritional status. Additionally, CT, MRI, endoscopy, and upper GI series examinations may be used to track and assist in analyzing the causes of postoperative complications.

Statistical Analysis The study will analyze the surgical prognosis, care priorities, common complications, and the management and outcomes of the hospital team for ESRD patients undergoing pancreatic surgery, aiming to provide diverse and specific treatment recommendations in the future.

Confidentiality and Privacy Protection To ensure patient privacy and personal information security, after querying the relevant data of enrolled subjects, the data sheet will use new codes to represent the subjects' identities. Experimenters and analysts will only have access to this de-linked data sheet for analysis. All electronic data will be password-protected and accessible only by specific personnel related to this project.

All data not used or after analysis will be stored at the NTU Department of Surgery for 15 years and then destroyed by shredder or incineration to remove identifiable personal data, unless required for medical or research purposes. Researchers (including external personnel) will sign a written pledge stating that medical record data will not be reused, disclosed to third parties, or used for purposes outside this study, unless required by law or audited by the Research Ethics Committee. If researchers encounter data that cannot directly identify identity, they will not attempt to identify individual patients. Collaborating external academic institutions or manufacturers must sign a research collaboration agreement.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males or females aged between 20 and 75 years. 2. Patients scheduled to undergo pancreatic surgery.

Exclusion Criteria:

* Patients under 20 or over 75 years of age at this hospital. 2. Presence of other active malignancies prior to diagnosis. 3. Minors, pregnant women, breastfeeding women, and patients with psychiatric disorders.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage renal disease and need pancreatic surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically relevant POPF and Clavian Dindo IIIA or higher complication | within 6 months after operation

IPD SHARING:
Plan to Share IPD: Undecided